CLINICAL TRIAL: NCT05923957
Title: The Impact of High Frequency Electrical Nerve Stimulation and Chiropractic Care on Sciatic Axonal Lesion Presenting as Painful Leg: Case Report
Status: Completed | Type: Observational
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Mshari Saleh Alghadier, Assistant Professor, Prince Sattam Bin Abdulaziz University
Other Study IDs: P.T-IMG-02/2023/507
Record Dates: First submitted 2023-06-09; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Sciatica Pain
Keywords: High frequency electrical stimulation; lumber spine; sciatic nerve; painful leg; gait training; chiropractic
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation; Exercise

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: High frequency electrical stimulation was done for thirty minutes per day for five days a week for four consecutive weeks. The stimulator provides a biphasic current of 100 Hz frequency. The pulse duration was 200 msec with an (on-off). Stimulus mode (20sec stimulation, 20 sec pause). The maximal stimulation amplitude was 40 - 60 mA
  Interventions: Other: TENS and Exercise

INTERVENTIONS:
Other: TENS and Exercise — High frequency electrical stimulation was done for thirty minutes per day for five days a week for four consecutive weeks. The stimulator provides a biphasic current of 100 Hz frequency. The pulse duration was 200 msec with an (on-off). Stimulus mode (20sec stimulation, 20 sec pause). The maximal stimulation amplitude was 40 - 60 mA

SUMMARY:
To present an evidence-based case report on the prognosis of a pediatric patient with right sciatica and painful leg. A 5-year-old girl with limping gait, presented with right-sided buttock and lower extremity pain and numbness. There has been a history of trauma prior to this 18-month ago. Following clinical examination, she was found to have numbness along the entire length of her right leg, in addition to a little sensory disturbance, accompanied by weakening in that leg. There was a generalized loss in sensation to pinprick as well as light touch, but it was most noticeable above the right knee joint. The remaining of the clinical exam was normal.

High frequency electrical stimulation was done for thirty minutes per day for five days a week for four consecutive weeks. The stimulator provides a biphasic current of 100 Hz frequency. The pulse duration was 200 msec with an (on-off). Stimulus mode (20sec stimulation, 20 sec pause). The maximal stimulation amplitude was 40 - 60 mA.

DETAILED DESCRIPTION:
A 5-year-old girl with limping gait, presented with right-sided buttock and lower extremity pain and numbness. There was a history of trauma preceding this eighteen months ago. There was diffuse decreased sensation to pinprick and light touch but mainly from above the right knee joint. The rest of the clinical examination was normal. The patient attended 20 sessions, which were structured to include High-frequency transcutaneous neuromuscular electrical nerve stimulation (TENS), chiropractic care, strengthening exercise for hamstring and back muscle and gait training (figure 1). Electrical stimulation was performed for 30 min /day for five days a week for four consecutive weeks, 100 Hz frequency with pulse duration 200 m sec with an (on-off) (20 sec stimulation, 20 sec pause) and maximum amplitude 40 - 60 mA. Two electrodes were placed on the back at the level of L5, S1 lumber spine and the other two electrodes were placed along the course of sciatic nerve on the back of the thigh. Chiropractic treatment sessions (manual manipulation refers to a high-velocity, short lever arm thrust that is applied to abnormal vertebra with the goal of improving functionality, reducing nerve irritability and restoring range of motion in the back) were scheduled for one month with frequency 5 sessions per week. strengthening program was three sets, ten repetitions and rest period of 1-2 minutes for low intensity or low repetition activity started by 2-3 days a week, then increase to 3-5 days a week as the strength progresses, amount of resistance 40%-60% of one-repetition maximum (1 RM). Mirror imaging and verbal promoting, Balance training and coordination to encourage normal gait.

EMG examination using concentric needle electrodes was carried bilaterally for the vastus medialis, tibialis anterior, extensor digitorum brevis and abductor halluces muscles and the right biceps femoris muscle. Motor conduction studies were carried out for both common peroneal, tibial and right main trunk of the right sciatic nerve.

ELIGIBILITY:
Inclusion Criteria:

* Sciatica nerve pain
* Able to attend 20 sessions
* Children age 5-10 years

Exclusion Criteria:

* Chronic pain
* Pain in the spine other than Sciatica

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with sciatica nerve pain
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Nerve conduction velocity | 4 weeks
  Motor conduction studies were carried out for both common peroneal, tibial and right main trunk of the right sciatic nerve.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the publication will be shared.
Supporting Information: CSR
Time Frame: 01/07/2023 - 01/07/2024
Access Criteria: Team researchers

REFERENCES:
- [Background] Vance CG, Rakel BA, Blodgett NP, DeSantana JM, Amendola A, Zimmerman MB, Walsh DM, Sluka KA. Effects of transcutaneous electrical nerve stimulation on pain, pain sensitivity, and function in people with knee osteoarthritis: a randomized controlled trial. Phys Ther. 2012 Jul;92(7):898-910. doi: 10.2522/ptj.20110183. Epub 2012 Mar 30. PMID 22466027
- [Background] Gordon T, Sulaiman O, Boyd JG. Experimental strategies to promote functional recovery after peripheral nerve injuries. J Peripher Nerv Syst. 2003 Dec;8(4):236-50. doi: 10.1111/j.1085-9489.2003.03029.x. PMID 14641648
- [Background] Kao CH, Chen JJ, Hsu YM, Bau DT, Yao CH, Chen YS. High-frequency electrical stimulation can be a complementary therapy to promote nerve regeneration in diabetic rats. PLoS One. 2013 Nov 12;8(11):e79078. doi: 10.1371/journal.pone.0079078. eCollection 2013. PMID 24265744
- [Background] Willand MP. Electrical Stimulation Enhances Reinnervation After Nerve Injury. Eur J Transl Myol. 2015 Aug 24;25(4):243-8. doi: 10.4081/ejtm.2015.5243. eCollection 2015 Aug 24. PMID 26913163
- [Background] Su HL, Chiang CY, Lu ZH, Cheng FC, Chen CJ, Sheu ML, Sheehan J, Pan HC. Late administration of high-frequency electrical stimulation increases nerve regeneration without aggravating neuropathic pain in a nerve crush injury. BMC Neurosci. 2018 Jun 25;19(1):37. doi: 10.1186/s12868-018-0437-9. PMID 29940857
- [Background] Baptista AF, Gomes JR, Oliveira JT, Santos SM, Vannier-Santos MA, Martinez AM. High- and low-frequency transcutaneous electrical nerve stimulation delay sciatic nerve regeneration after crush lesion in the mouse. J Peripher Nerv Syst. 2008 Mar;13(1):71-80. doi: 10.1111/j.1529-8027.2008.00160.x. PMID 18346233
- [Background] Alrashdan MS, Park JC, Sung MA, Yoo SB, Jahng JW, Lee TH, Kim SJ, Lee JH. Thirty minutes of low intensity electrical stimulation promotes nerve regeneration after sciatic nerve crush injury in a rat model. Acta Neurol Belg. 2010 Jun;110(2):168-79. PMID 20873447
- [Background] Teodori RM, Silva AM, Silva MT, Oliveira LS, Polacow ML, Guirro EC. High-voltage electrical stimulation improves nerve regeneration after sciatic crush injury. Rev Bras Fisioter. 2011 Aug-Sep;15(4):325-31. doi: 10.1590/s1413-35552011005000008. Epub 2011 Aug 5. PMID 21975682
- [Background] Foecking EM, Fargo KN, Coughlin LM, Kim JT, Marzo SJ, Jones KJ. Single session of brief electrical stimulation immediately following crush injury enhances functional recovery of rat facial nerve. J Rehabil Res Dev. 2012;49(3):451-8. doi: 10.1682/jrrd.2011.03.0033. PMID 22773203
- [Background] Bowman BR, McNeal DR. Response of single alpha motoneurons to high-frequency pulse trains. Firing behavior and conduction block phenomenon. Appl Neurophysiol. 1986;49(3):121-38. doi: 10.1159/000100137. PMID 3827239
- [Background] WOO MY, CAMPBELL B. ASYNCHRONOUS FIRING AND BLOCK OF PERIPHERAL NERVE CONDUCTION BY 20 KC ALTERNATING CURRENT. Bull Los Angel Neuro Soc. 1964 Jun;29:87-94. No abstract available. PMID 14169956
- [Background] TANNER JA. Reversible blocking of nerve conduction by alternating-current excitation. Nature. 1962 Aug 18;195:712-3. doi: 10.1038/195712b0. No abstract available. PMID 13919574
- [Background] Porcino A, Solomonian L, Zylich S, Gluvic B, Doucet C, Vohra S. Pediatric training and practice of Canadian chiropractic and naturopathic doctors: a 2004-2014 comparative study. BMC Complement Altern Med. 2017 Dec 1;17(1):512. doi: 10.1186/s12906-017-2024-5. PMID 29191235
- [Background] Donnelly C, Stegmuller J, Blazevich AJ, Crettaz von Roten F, Kayser B, Neyroud D, Place N. Modulation of torque evoked by wide-pulse, high-frequency neuromuscular electrical stimulation and the potential implications for rehabilitation and training. Sci Rep. 2021 Mar 18;11(1):6399. doi: 10.1038/s41598-021-85645-0. PMID 33737664
- [Background] Kilgore KL, Bhadra N. Nerve conduction block utilising high-frequency alternating current. Med Biol Eng Comput. 2004 May;42(3):394-406. doi: 10.1007/BF02344716. PMID 15191086
- [Background] Egginton S, Hudlicka O. Early changes in performance, blood flow and capillary fine structure in rat fast muscles induced by electrical stimulation. J Physiol. 1999 Feb 15;515 ( Pt 1)(Pt 1):265-75. doi: 10.1111/j.1469-7793.1999.265ad.x. PMID 9925896
- [Background] 2. Katirji B, editor. 2002. Compressive and entrapment neuropathies of the lower extremity in Neuromuscular Disorders in Clinical Practice. Boston: Butterworth Heinemann;. p. 787-96.
- [Background] Distad BJ, Weiss MD. Clinical and electrodiagnostic features of sciatic neuropathies. Phys Med Rehabil Clin N Am. 2013 Feb;24(1):107-20. doi: 10.1016/j.pmr.2012.08.023. Epub 2012 Oct 31. PMID 23177034